CLINICAL TRIAL: NCT03750240
Title: Metabolic Sodium MRI to Assess Early Response of Breast Cancer to Neoadjuvant Chemotherapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: technical difficulties for scans on the research MRI system
Sponsor: NYU Langone Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-00269
Record Dates: First submitted 2018-11-20; First posted 2018-11-21 (Actual); Results first posted 2022-08-24 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Breast Cancer; Triple Negative Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Triple Negative Breast Cancer Patients (Experimental): scanned 4 times to assess breast cancer response to NACT with the proposed method.
  Interventions: Diagnostic Test: Sodium (Na) Magnetic Resonance Imaging (MRI); Diagnostic Test: Dynamic Contrast- Enhanced (DCE) MRI

INTERVENTIONS:
Diagnostic Test: Sodium (Na) Magnetic Resonance Imaging (MRI) — Two Na data will be acquired:
  1. FLORET without Inversion Recovery (IR), and
  2. FLORET with IR
Diagnostic Test: Dynamic Contrast- Enhanced (DCE) MRI — DCE MRI will be acquired subsequent to Na MRI to prevent influence of the contrast agent on 23 Na data

SUMMARY:
Neoadjuvant chemotherapy (NACT) is administered to treat invasive breast cancer before surgery. It offers the opportunity to evaluate tumor response to treatment in aggressive disease, and guide additional therapies for patients with inadequate response, if detected early. Investigators propose to develop a sodium breast MRI technique that will allow to assess the early metabolic response of breast cancer to NACT, occurring before late structural changes can be detected with standard MRI.

This study will scan 12 patients using 1H/23Na MRI at 7 T and DCE MRI with triple-negative breast cancer undergoing AC-T therapy (2 months of Adriamycin + Cyclophosphamide, then 3 months of Taxol): at baseline (pre-NACT); after the first AC cycle (2 weeks); after AC treatment (2 months); after complete NACT (5 months, pre-surgery).

ELIGIBILITY:
Inclusion Criteria:

* Women with no sign of breast cancer as controls
* Non-pregnant and non-lactating
* Ability to understand and willingness to sign a written consent

Exclusion Criteria:

* Contra-indications to MRI (i.e., ferromagnetic prostheses, metallic surgical implants that are not compatible with an MRI machine, claustrophobia etc.)
* Medical condition such as uncontrolled infection (including HIV), uncontrolled diabetes mellitus or cardiac disease which, in the opinion of the treating physician, would make this protocol unreasonably hazardous for the patient.
* Pregnant or lactating women, women using hormonal treatment in the 6 months prior to the study.
* Women with history of breast disease, previous breast surgery, or breast implants.
* Patients with a currently active second malignancy other than non-melanoma skin cancers. Patients are not considered to have a currently active malignancy if they have completed therapy and are free of disease for 3 years.
* Psychiatric illness or other conditions and circumstances which could prevent the patient from being compliant with the protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 2 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2021-06-24 (Actual); Study Completion 2021-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Madelin, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Triple Negative Breast Cancer Patients: scanned 4 times to assess breast cancer response to NACT with the proposed method.
  Sodium (Na) Magnetic Resonance Imaging (MRI): Two Na data will be acquired:
  1. FLORET without Inversion Recovery (IR), and
  2. FLORET with IR
  Dynamic Contrast- Enhanced (DCE) MRI: DCE MRI will be acquired subsequent to Na MRI to prevent influence of the contrast agent on 23 Na data
Period: Overall Study
Arm/Group | Triple Negative Breast Cancer Patients
Started | 2
Completed | 0
Not Completed | 2
Not completed — Technical Difficulties | 2

BASELINE CHARACTERISTICS:
Arm/Group | Triple Negative Breast Cancer Patients
Number analyzed (Participants) | 2
Age, Continuous [Mean (Full Range); unit: years] | 54.5 [51 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Tumor Size
Description: Dynamic contrast-enhanced MRI will be used to measure tumor size before and after treatment.
Time Frame: Baseline, 2 Years
Population: The study was terminated due to technical difficulties; therefore, no follow-ups during or after therapy were performed with only scans at baseline
Arm/Group | Triple Negative Breast Cancer Patients
Number analyzed (Participants) | 0

2. Secondary Outcome: Total Sodium Concentration (TSC)
Description: TSC was directly measured from 23Na images using a phantom calibration
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mM
Arm/Group | Triple Negative Breast Cancer Patients
Number analyzed (Participants) | 2
mM
  Participant 1 | 47.0 (11.1)
  Participant 2 | 39.2 (15.2)

3. Secondary Outcome: Intracellular Sodium Concentration (CIC)
Description: CIC is derived from this equation: TSC = ECV · CEC + ICV · CIC + (1 -WF) · Cfat
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mM
Arm/Group | Triple Negative Breast Cancer Patients
Number analyzed (Participants) | 2
mM
  Participant 1 | 29.6 (17.9)
  Participant 2 | 27.2 (21.1)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Triple Negative Breast Cancer Patients
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-02): https://cdn.clinicaltrials.gov/large-docs/40/NCT03750240/Prot_SAP_000.pdf